CLINICAL TRIAL: NCT01846455
Title: Pharmacokinetics of Buprenorphine and Naloxone in Subjects With Mild to Severe Hepatic Impairment (Child-Pugh Classes, A, B, and C), in HCV-Seropositive Subjects, and in Healthy Volunteers
Brief Title: Single Dose Pharmacokinetics of Suboxone Study in Hepatic Impaired Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RB-US-08-0003
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Results first posted 2016-10-24 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-09

CONDITIONS: Hepatic Failure; Hepatic Impairment; Chronic Hepatitis C Infection With Hepatic Coma
Keywords: Hepatic; Hepatitis C Virus; Suboxone; Buprenorphine; Naloxone
MeSH Terms: conditions — Liver Failure; Hepatitis C | interventions — Buprenorphine, Naloxone Drug Combination; Promethazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Hepatic Impairment: Child-Pugh A (Experimental): Participants with chronic liver disease and classified as Child-Pugh Grade A had a score of 5-6 (out of 15) which correlates with a good prognosis. Each participant received one sublingual tablet of Suboxone® (2mg buprenorphine with 0.5 mg naloxone) on Day 1.
  Interventions: Drug: 2.0mg Buprenorphine/0.5mg Naloxone; Drug: Promethazine
- Hepatic Impairment: Child-Pugh B (Experimental): Participants with chronic liver disease and classified as Child-Pugh Grade B had a score of 7-9 (out of 15) which correlates with significant functional liver compromise. Each participant received one sublingual tablet of Suboxone® (2mg buprenorphine with 0.5 mg naloxone) on Day 1.
  Interventions: Drug: 2.0mg Buprenorphine/0.5mg Naloxone; Drug: Promethazine
- Hepatic Impairment: Child-Pugh C (Experimental): Participants with chronic liver disease and classified as Child-Pugh Grade C had a score of 10-15 (out of 15) which correlates with decompensated liver disease. Each participant received one sublingual tablet of Suboxone® (2mg buprenorphine with 0.5 mg naloxone) on Day 1.
  Interventions: Drug: 2.0mg Buprenorphine/0.5mg Naloxone; Drug: Promethazine
- HCV Without Hepatic Impairment (Experimental): Participants with hepatitis C virus (HCV) without hepatic impairment received one sublingual tablet of Suboxone® (2mg buprenorphine with 0.5 mg naloxone) on Day 1.
  Interventions: Drug: 2.0mg Buprenorphine/0.5mg Naloxone; Drug: Promethazine
- No Hepatic Disease or Impairment (Active Comparator): Participants with no hepatic disease or impairment received one sublingual tablet of Suboxone® (2mg buprenorphine with 0.5 mg naloxone) on Day 1.
  Interventions: Drug: 2.0mg Buprenorphine/0.5mg Naloxone; Drug: Promethazine

INTERVENTIONS:
Drug: 2.0mg Buprenorphine/0.5mg Naloxone — Each participant received a single sublingual dose of Suboxone® on Day 1 following a fast of at least 8 hours prior to dosing and 2 hours after dosing.
  Other Names: Suboxone®
Drug: Promethazine — Each participant received a 25-mg or 50-mg promethazine oral dose 30 minutes before Suboxone® administration and then 25-mg promethazine orally or by rectal suppositories every 4 hours as needed for nausea and vomiting during the first 48 hours after Suboxone® administration.

SUMMARY:
The objective was to determine if hepatitis C virus (HCV) infection or mild to severe hepatic impairment (Child-Pugh Classes A, B, and C) altered the PK of buprenorphine, norbuprenorphine, or naloxone.

DETAILED DESCRIPTION:
This will be a multi-center, open-label study. After providing informed consent, subjects will undergo an outpatient screening period of up to 21 days. Screening procedures will include an assessment of mental status which will be repeated before dosing. Eligible subjects will then undergo hospital intake procedures and reside at the investigational site until Day 5. Subjects will be enrolled in 5-treatment groups as follows: (1) Group 1: Subjects with hepatic impairment classified as Child-Pugh A; (2) Group 2: Subjects with hepatic impairment classified as Child-Pugh B; (3) Group 3: Subjects with hepatic impairment classified as Child-Pugh C; (4) Group 4: Subjects with Hepatitis C Virus (HCV) infection but without hepatic impairment; and (5) Group 5: Subjects without hepatic disease or impairment. Group 5 is used as a control group

ELIGIBILITY:
Inclusion Criteria:

* Males or females between the ages of 18 and 65 years, inclusive
* Females should be surgically sterile, 2 years post-menopausal or have a negative plasma β-human chorionic gonadotropin (β-hCG) pregnancy test. Subjects of child-bearing potential must take reasonable precautions during the study to avoid pregnancy by agreeing to remain abstinent or to practice double-barrier forms of birth control from the time of informed consent through the last study visit. A negative plasma pregnancy (β-hCG) test at Screening and upon admission to the investigational site. Testing for β-hCG will need to be timed to ensure a negative pregnancy result at Day 1.
* Male subject agrees to use barrier contraception and spermicide when engaging in sexual activity with a female of child-bearing potential for at least 28 days after the study medication dose.
* Male subject agrees to refrain from sperm donations for the entire duration of the study and for at least 90 days after the study drug dose.
* Body mass index (BMI) of ≥ 18 to ≤ 33 kg^m2.
* Subject agrees to the conditions of the study and signs the informed consent form

Exclusion Criteria:

* Medical conditions: (a) pregnancy; and (b) breastfeeding
* Psychiatric conditions: (a) current treatment for opioid addiction with substitution therapies; (b) active history of bipolar I, bipolar II, schizophrenia, schizophreniform; schizoaffective; mania, hypomania, or severe post-traumatic stress disorder; and (c) presence of suicidal behavior within the year before informed consent or suicidal intent within the 30 days before informed consent as documented by the Columbia Suicide Severity Rating Scale
* Hypersensitivity to opioids, defined as intractable vomiting, severe constipation, or severe pruritus after opioid treatment
* Subject has a known intolerance or hypersensitivity to buprenorphine or naloxone or any excipients in the Suboxone tablet formulation
* In the judgment of the investigator, any other condition that would preclude safe, useful, or consistent participation in the study
* Use of any investigational medication or investigational medical device in the 30 days before informed consent
* Hepatic encephalopathy greater than West Haven Grade 2
* Donation of > 250 ml of blood within previous 30 days
* Systolic BP ≤ 90 or ≥ 160 mmHg and/or Diastolic BP < 60 mmHg or > 100 mmHg
* History of cholecystectomy
* History or current acquired immunodeficiency syndrome (AIDS) or human immunodeficiency virus (HIV) antibodies
* Estimated creatinine clearance rate (eC Cr) using Cockcroft-Gault formula < 60 mL/min
* More than 1 missed appointment during Screening
* Currently under mandate by the criminal justice system or Child and Family Services to participate in drug abuse treatment
* Participation in drug or alcohol dependence treatment in the 30 days before informed consent
* Positive urine drug screen result for amphetamines, methamphetamine, barbiturates, benzodiazepines, buprenorphine, cannabinoids, cocaine, methadone, opioids, oxycodone, or phencyclidine which, in the judgment of the investigator, is indicative of non-prescribed drug use; and/or positive urine alcohol screen result in which, in the judgment of the investigator, is indicative of alcohol abuse or alcoholism
* Consumption of prohibited medications within 1 week of informed consent, including buprenorphine
* Consumption of grapefruit and grapefruit juice for at least one week before the study dose and until the end of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2012-09; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lasseter, MD, Principal Investigator — Clinical Pharmacology of Miami, Inc.; Thomas Marabury, MD, Principal Investigator — Orlando Clinical Research Center; Eric J. Lawitz, MD, Principal Investigator — American Research Corporation (ARC)
Locations (3):
- United States (3):
  - Clinical Pharmacology of Miami, Inc., Hialeah, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - American Research Corporation (ARC), San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nasser AF, Heidbreder C, Liu Y, Fudala PJ. Pharmacokinetics of Sublingual Buprenorphine and Naloxone in Subjects with Mild to Severe Hepatic Impairment (Child-Pugh Classes A, B, and C), in Hepatitis C Virus-Seropositive Subjects, and in Healthy Volunteers. Clin Pharmacokinet. 2015 Aug;54(8):837-49. doi: 10.1007/s40262-015-0238-6. PMID 25603822

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hepatic Impairment: Child-Pugh A | Hepatic Impairment: Child-Pugh B | Hepatic Impairment: Child-Pugh C | HCV Without Hepatic Impairment | No Hepatic Disease or Impairment
Started | 9 | 8 | 8 | 10 | 8
PK Population | 6 | 7 | 6 | 6 | 8
Completed | 9 | 8 | 8 | 10 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Total: Total of all reporting groups
Arm/Group | Hepatic Impairment: Child-Pugh A | Hepatic Impairment: Child-Pugh B | Hepatic Impairment: Child-Pugh C | HCV Without Hepatic Impairment | No Hepatic Disease or Impairment | Total
Number analyzed (Participants) | 9 | 8 | 8 | 10 | 8 | 43
Age, Continuous [Mean (Full Range); unit: years] | 58.0 [51 to 62] | 58.6 [52 to 63] | 53.9 [42 to 65] | 53.0 [43 to 59] | 57.1 [49 to 62] | 56.0 [42 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 1 | 6 | 4 | 18
  Male | 6 | 4 | 7 | 4 | 4 | 25
Race/Ethnicity, Customized [Number; unit: participants]
  White | 6 | 7 | 8 | 8 | 7 | 36
  Black or African American | 2 | 1 | 0 | 1 | 1 | 5
  Asian | 1 | 0 | 0 | 1 | 0 | 2
Weight [Mean (Full Range); unit: kg] | 74.2 [54.0 to 92.5] | 75.4 [56.0 to 95.0] | 82.2 [64.8 to 103.0] | 74.7 [60.2 to 109.0] | 76.6 [69.2 to 83.6] | 76.5 [54.0 to 109.0]
Body Mass Index [Mean (Full Range); unit: kg/m^2] | 25.5 [18.7 to 32.8] | 27.0 [20.3 to 32.3] | 27.9 [23.2 to 32.8] | 26.2 [20.6 to 32.9] | 29.3 [22.1 to 32.2] | 27.1 [18.7 to 32.9]

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration (AUC0-last) of Buprenorphine, Norbuprenorphine, Naloxone and Naloxone-3-β-D-Glucuronide
Description: AUC0-last was calculated for buprenorphine, norbuprenorphine, naloxone, and naloxone-3-β-D-glucuronide using non-compartmental analysis:
  AUC0-last = AUC from time 0 to the time of the last measurable plasma concentration, calculated using the linear trapezoidal rule.
Time Frame: before dosing (time 0; Baseline) and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144, and 168 hours after dosing
Population: The PK population included participants without any major protocol deviations who contributed PK samples and had sufficient evaluable data for the calculation of PK parameters. Eight enrolled participants were excluded due to emesis observed within 4 hours postdose, and two due to protocol violations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Hepatic Impairment: Child-Pugh A | Hepatic Impairment: Child-Pugh B | Hepatic Impairment: Child-Pugh C | HCV Without Hepatic Impairment | No Hepatic Disease or Impairment
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 8
ng*hr/mL
  Buprenorphine | 8.89 (33.3) | 14.7 (55.0) | 25.2 (53.7) | 7.02 (36.5) | 8.95 (49.4)
  Norbuprenorphine | 12.5 (119) | 9.51 (71.4) | 2.25 (118) | 9.91 (43.4) | 15.0 (51.8)
  Naloxone | 0.0726 (41.8) | 0.291 (195) | 1.28 (60.2) | 0.0968 (73.0) | 0.0915 (50.9)
  Naloxone-3-β-D-Glucuronide | 19.3 (31.9) | 27.9 (33.6) | 20.6 (40.2) | 19.1 (21.8) | 22.5 (15.8)
Statistical Analysis 1: Comparison: Hepatic Impairment: Child-Pugh A vs No Hepatic Disease or Impairment; Buprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 99.34, 90% CI 2-sided [66.05 to 149.43]
Statistical Analysis 2: Comparison: Hepatic Impairment: Child-Pugh B vs No Hepatic Disease or Impairment; Buprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 163.88, 90% CI 2-sided [110.82 to 242.34]
Statistical Analysis 3: Comparison: Hepatic Impairment: Child-Pugh C vs No Hepatic Disease or Impairment; Buprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 281.43, 90% CI 2-sided [187.10 to 423.33]
Statistical Analysis 4: Comparison: HCV Without Hepatic Impairment vs No Hepatic Disease or Impairment; Buprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 78.43, 90% CI 2-sided [52.14 to 117.98]
Statistical Analysis 5: Comparison: Hepatic Impairment: Child-Pugh A vs HCV Without Hepatic Impairment; Buprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 126.66, 90% CI 2-sided [81.87 to 195.97]
Statistical Analysis 6: Comparison: Hepatic Impairment: Child-Pugh B vs HCV Without Hepatic Impairment; Buprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 208.94, 90% CI 2-sided [137.21 to 318.18]
Statistical Analysis 7: Comparison: Hepatic Impairment: Child-Pugh C vs HCV Without Hepatic Impairment; Buprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 358.83, 90% CI 2-sided [231.92 to 555.17]
Statistical Analysis 8: Comparison: Hepatic Impairment: Child-Pugh A vs No Hepatic Disease or Impairment; Norbuprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 78.09, 90% CI 2-sided [44.03 to 138.49]
Statistical Analysis 9: Comparison: Hepatic Impairment: Child-Pugh B vs No Hepatic Disease or Impairment; Norbuprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 74.78, 90% CI 2-sided [39.26 to 142.41]
Statistical Analysis 10: Comparison: Hepatic Impairment: Child-Pugh C vs No Hepatic Disease or Impairment; Norbuprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 11.45, 90% CI 2-sided [6.35 to 20.66]
Statistical Analysis 11: Comparison: HCV Without Hepatic Impairment vs No Hepatic Disease or Impairment; Norbuprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 71.08, 90% CI 2-sided [39.00 to 129.49]
Statistical Analysis 12: Comparison: Hepatic Impairment: Child-Pugh A vs HCV Without Hepatic Impairment; Norbuprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 109.90, 90% CI 2-sided [58.14 to 207.75]
Statistical Analysis 13: Comparison: Hepatic Impairment: Child-Pugh B vs HCV Without Hepatic Impairment; Norbuprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 105.23, 90% CI 2-sided [52.17 to 212.24]
Statistical Analysis 14: Comparison: Hepatic Impairment: Child-Pugh C vs HCV Without Hepatic Impairment; Norbuprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 16.12, 90% CI 2-sided [8.40 to 30.94]
Statistical Analysis 15: Comparison: Hepatic Impairment: Child-Pugh A vs No Hepatic Disease or Impairment; Naloxone; Test type: Superiority or Other; ratio of parameter means, % = 79.30, 90% CI 2-sided [40.03 to 157.12]
Statistical Analysis 16: Comparison: Hepatic Impairment: Child-Pugh B vs No Hepatic Disease or Impairment; Naloxone; Test type: Superiority or Other; ratio of parameter means, % = 317.58, 90% CI 2-sided [164.93 to 611.54]
Statistical Analysis 17: Comparison: Hepatic Impairment: Child-Pugh C vs No Hepatic Disease or Impairment; Naloxone; Test type: Superiority or Other; ratio of parameter means, % = 1401.85, 90% CI 2-sided [707.55 to 2777.46]
Statistical Analysis 18: Comparison: HCV Without Hepatic Impairment vs No Hepatic Disease or Impairment; Naloxone; Test type: Superiority or Other; ratio of parameter means, % = 105.78, 90% CI 2-sided [53.39 to 209.59]
Statistical Analysis 19: Comparison: Hepatic Impairment: Child-Pugh A vs HCV Without Hepatic Impairment; Naloxone; Test type: Superiority or Other; ratio of parameter means, % = 74.97, 90% CI 2-sided [36.09 to 155.71]
Statistical Analysis 20: Comparison: Hepatic Impairment: Child-Pugh B vs HCV Without Hepatic Impairment; Naloxone; Test type: Superiority or Other; ratio of parameter means, % = 300.22, 90% CI 2-sided [148.44 to 607.21]
Statistical Analysis 21: Comparison: Hepatic Impairment: Child-Pugh C vs HCV Without Hepatic Impairment; Naloxone; Test type: Superiority or Other; ratio of parameter means, % = 1325.22, 90% CI 2-sided [638.03 to 2752.55]
Statistical Analysis 22: Comparison: Hepatic Impairment: Child-Pugh A vs No Hepatic Disease or Impairment; Naloxone-3-β-D-Glucuronide; Test type: Superiority or Other; ratio of parameter means, % = 85.87, 90% CI 2-sided [66.06 to 111.61]
Statistical Analysis 23: Comparison: Hepatic Impairment: Child-Pugh B vs No Hepatic Disease or Impairment; Naloxone-3-β-D-Glucuronide; Test type: Superiority or Other; ratio of parameter means, % = 123.77, 90% CI 2-sided [96.27 to 159.13]
Statistical Analysis 24: Comparison: Hepatic Impairment: Child-Pugh C vs No Hepatic Disease or Impairment; Naloxone-3-β-D-Glucuronide; Test type: Superiority or Other; ratio of parameter means, % = 91.26, 90% CI 2-sided [70.21 to 118.62]
Statistical Analysis 25: Comparison: HCV Without Hepatic Impairment vs No Hepatic Disease or Impairment; Naloxone-3-β-D-Glucuronide; Test type: Superiority or Other; ratio of parameter means, % = 84.78, 90% CI 2-sided [65.23 to 110.20]
Statistical Analysis 26: Comparison: Hepatic Impairment: Child-Pugh A vs HCV Without Hepatic Impairment; Naloxone-3-β-D-Glucuronide; Test type: Superiority or Other; ratio of parameter means, % = 101.28, 90% CI 2-sided [76.52 to 134.06]
Statistical Analysis 27: Comparison: Hepatic Impairment: Child-Pugh B vs HCV Without Hepatic Impairment; Naloxone-3-β-D-Glucuronide; Test type: Superiority or Other; ratio of parameter means, % = 145.99, 90% CI 2-sided [111.43 to 191.26]
Statistical Analysis 28: Comparison: Hepatic Impairment: Child-Pugh C vs HCV Without Hepatic Impairment; Naloxone-3-β-D-Glucuronide; Test type: Superiority or Other; ratio of parameter means, % = 107.64, 90% CI 2-sided [81.33 to 142.47]

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Buprenorphine, Norbuprenorphine, Naloxone and Naloxone-3-β-D-Glucuronide
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Hepatic Impairment: Child-Pugh A | Hepatic Impairment: Child-Pugh B | Hepatic Impairment: Child-Pugh C | HCV Without Hepatic Impairment | No Hepatic Disease or Impairment
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 8
ng/mL
  Buprenorphine | 1.10 (52.2) | 1.04 (46.5) | 1.40 (27.4) | 0.933 (30.5) | 0.913 (53.2)
  Norbuprenorphine | 0.358 (99.0) | 0.180 (73.2) | 0.128 (60.6) | 0.203 (61.0) | 0.265 (59.8)
  Naloxone | 0.0287 (62.7) | 0.0773 (159) | 0.323 (28.7) | 0.0361 (83.8) | 0.0286 (68.1)
  Naloxone-3-β-D-Glucuronide | 9.02 (29.8) | 9.03 (21.8) | 6.75 (40.0) | 6.80 (14.7) | 8.12 (30.5)
Statistical Analysis 1: Comparison: Hepatic Impairment: Child-Pugh A vs No Hepatic Disease or Impairment; Buprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 120.02, 90% CI 2-sided [83.35 to 172.82]
Statistical Analysis 2: Comparison: Hepatic Impairment: Child-Pugh B vs No Hepatic Disease or Impairment; Buprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 107.85, 90% CI 2-sided [75.85 to 153.36]
Statistical Analysis 3: Comparison: Hepatic Impairment: Child-Pugh C vs No Hepatic Disease or Impairment; Buprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 171.76, 90% CI 2-sided [117.93 to 250.15]
Statistical Analysis 4: Comparison: HCV Without Hepatic Impairment vs No Hepatic Disease or Impairment; Buprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 112.82, 90% CI 2-sided [77.66 to 163.91]
Statistical Analysis 5: Comparison: Hepatic Impairment: Child-Pugh A vs HCV Without Hepatic Impairment; Buprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 106.38, 90% CI 2-sided [71.43 to 158.43]
Statistical Analysis 6: Comparison: Hepatic Impairment: Child-Pugh B vs HCV Without Hepatic Impairment; Buprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 95.59, 90% CI 2-sided [64.36 to 141.99]
Statistical Analysis 7: Comparison: Hepatic Impairment: Child-Pugh C vs HCV Without Hepatic Impairment; Buprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 152.24, 90% CI 2-sided [103.08 to 224.83]
Statistical Analysis 8: Comparison: Hepatic Impairment: Child-Pugh A vs No Hepatic Disease or Impairment; Norbuprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 135.17, 90% CI 2-sided [75.44 to 242.16]
Statistical Analysis 9: Comparison: Hepatic Impairment: Child-Pugh B vs No Hepatic Disease or Impairment; Norbuprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 67.87, 90% CI 2-sided [38.82 to 118.68]
Statistical Analysis 10: Comparison: Hepatic Impairment: Child-Pugh C vs No Hepatic Disease or Impairment; Norbuprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 48.39, 90% CI 2-sided [27.01 to 86.69]
Statistical Analysis 11: Comparison: HCV Without Hepatic Impairment vs No Hepatic Disease or Impairment; Norbuprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 76.59, 90% CI 2-sided [42.75 to 137.22]
Statistical Analysis 12: Comparison: Hepatic Impairment: Child-Pugh A vs HCV Without Hepatic Impairment; Norbuprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 176.48, 90% CI 2-sided [94.62 to 329.17]
Statistical Analysis 13: Comparison: Hepatic Impairment: Child-Pugh B vs HCV Without Hepatic Impairment; Norbuprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 88.62, 90% CI 2-sided [48.60 to 161.59]
Statistical Analysis 14: Comparison: Hepatic Impairment: Child-Pugh C vs HCV Without Hepatic Impairment; Norbuprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 63.17, 90% CI 2-sided [33.87 to 117.83]
Statistical Analysis 15: Comparison: Hepatic Impairment: Child-Pugh A vs No Hepatic Disease or Impairment; Naloxone; Test type: Superiority or Other; ratio of parameter means, % = 100.41, 90% CI 2-sided [51.30 to 196.53]
Statistical Analysis 16: Comparison: Hepatic Impairment: Child-Pugh B vs No Hepatic Disease or Impairment; Naloxone; Test type: Superiority or Other; ratio of parameter means, % = 270.00, 90% CI 2-sided [141.86 to 513.90]
Statistical Analysis 17: Comparison: Hepatic Impairment: Child-Pugh C vs No Hepatic Disease or Impairment; Naloxone; Test type: Superiority or Other; ratio of parameter means, % = 1129.81, 90% CI 2-sided [577.22 to 2211.44]
Statistical Analysis 18: Comparison: HCV Without Hepatic Impairment vs No Hepatic Disease or Impairment; Naloxone; Test type: Superiority or Other; ratio of parameter means, % = 126.25, 90% CI 2-sided [64.50 to 247.11]
Statistical Analysis 19: Comparison: Hepatic Impairment: Child-Pugh A vs HCV Without Hepatic Impairment; Naloxone; Test type: Superiority or Other; ratio of parameter means, % = 79.53, 90% CI 2-sided [38.79 to 163.06]
Statistical Analysis 20: Comparison: Hepatic Impairment: Child-Pugh B vs HCV Without Hepatic Impairment; Naloxone; Test type: Superiority or Other; ratio of parameter means, % = 213.86, 90% CI 2-sided [107.07 to 427.17]
Statistical Analysis 21: Comparison: Hepatic Impairment: Child-Pugh C vs HCV Without Hepatic Impairment; Naloxone; Test type: Superiority or Other; ratio of parameter means, % = 894.91, 90% CI 2-sided [436.49 to 1834.80]
Statistical Analysis 22: Comparison: Hepatic Impairment: Child-Pugh A vs No Hepatic Disease or Impairment; Naloxone-3-β-D-Glucuronide; Test type: Superiority or Other; ratio of parameter means, % = 111.03, 90% CI 2-sided [85.94 to 143.44]
Statistical Analysis 23: Comparison: Hepatic Impairment: Child-Pugh B vs No Hepatic Disease or Impairment; Naloxone-3-β-D-Glucuronide; Test type: Superiority or Other; ratio of parameter means, % = 111.22, 90% CI 2-sided [87.02 to 142.16]
Statistical Analysis 24: Comparison: Hepatic Impairment: Child-Pugh C vs No Hepatic Disease or Impairment; Naloxone-3-β-D-Glucuronide; Test type: Superiority or Other; ratio of parameter means, % = 83.09, 90% CI 2-sided [64.32 to 107.35]
Statistical Analysis 25: Comparison: HCV Without Hepatic Impairment vs No Hepatic Disease or Impairment; Naloxone-3-β-D-Glucuronide; Test type: Superiority or Other; ratio of parameter means, % = 83.66, 90% CI 2-sided [64.75 to 108.08]
Statistical Analysis 26: Comparison: Hepatic Impairment: Child-Pugh A vs HCV Without Hepatic Impairment; Naloxone-3-β-D-Glucuronide; Test type: Superiority or Other; ratio of parameter means, % = 132.72, 90% CI 2-sided [100.93 to 174.53]
Statistical Analysis 27: Comparison: Hepatic Impairment: Child-Pugh B vs HCV Without Hepatic Impairment; Naloxone-3-β-D-Glucuronide; Test type: Superiority or Other; ratio of parameter means, % = 132.95, 90% CI 2-sided [102.12 to 173.10]
Statistical Analysis 28: Comparison: Hepatic Impairment: Child-Pugh C vs HCV Without Hepatic Impairment; Naloxone-3-β-D-Glucuronide; Test type: Superiority or Other; ratio of parameter means, % = 99.33, 90% CI 2-sided [75.54 to 130.61]

3. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUC0-inf) of Buprenorphine, Norbuprenorphine, Naloxone and Naloxone-3-β-D-Glucuronide
Description: The extrapolation to infinity was done using the terminal phase.
  AUC0-inf = AUC0-last + Ct/λz
  Where Ct was the last observed quantifiable concentration and λz was the apparent terminal phase elimination rate constant.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Hepatic Impairment: Child-Pugh A | Hepatic Impairment: Child-Pugh B | Hepatic Impairment: Child-Pugh C | HCV Without Hepatic Impairment | No Hepatic Disease or Impairment
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 8
ng*hr/mL
  Buprenorphine (5,4,5,3,6) | 11.0 (30.8) | 18.9 (58.4) | 25.5 (44.6) | 8.61 (22.6) | 10.3 (56.0)
  Norbuprenorphine (3,3,1,3,3) | 25.4 (25.5) | 17.1 (77.4) | 6.67 (NA) — Value is for a single participant | 13.9 (58.6) | 16.0 (23.0)
  Naloxone (5,6,5,4,7) | 0.0671 (18.7) | 0.274 (195) | 1.45 (57.0) | 0.0851 (57.0) | 0.0971 (53.4)
  Naloxone-3-β-D-Glucuronide (5,7,6,5,4) | 21.9 (28.0) | 28.9 (32.7) | 21.3 (38.5) | 21.5 (15.0) | 26.0 (12.4)
Statistical Analysis 1: Comparison: Hepatic Impairment: Child-Pugh A vs No Hepatic Disease or Impairment; Buprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 125.19, 90% CI 2-sided [79.46 to 197.24]
Statistical Analysis 2: Comparison: Hepatic Impairment: Child-Pugh B vs No Hepatic Disease or Impairment; Buprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 220.97, 90% CI 2-sided [135.33 to 360.81]
Statistical Analysis 3: Comparison: Hepatic Impairment: Child-Pugh C vs No Hepatic Disease or Impairment; Buprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 249.28, 90% CI 2-sided [162.19 to 383.14]
Statistical Analysis 4: Comparison: HCV Without Hepatic Impairment vs No Hepatic Disease or Impairment; Buprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 94.44, 90% CI 2-sided [56.44 to 158.02]
Statistical Analysis 5: Comparison: Hepatic Impairment: Child-Pugh A vs HCV Without Hepatic Impairment; Buprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 132.57, 90% CI 2-sided [78.86 to 222.84]
Statistical Analysis 6: Comparison: Hepatic Impairment: Child-Pugh B vs HCV Without Hepatic Impairment; Buprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 233.99, 90% CI 2-sided [135.63 to 403.68]
Statistical Analysis 7: Comparison: Hepatic Impairment: Child-Pugh C vs HCV Without Hepatic Impairment; Buprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 263.97, 90% CI 2-sided [155.52 to 448.03]
Statistical Analysis 8: Comparison: Hepatic Impairment: Child-Pugh A vs No Hepatic Disease or Impairment; Norbuprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 159.38, 90% CI 2-sided [78.21 to 324.79]
Statistical Analysis 9: Comparison: Hepatic Impairment: Child-Pugh B vs No Hepatic Disease or Impairment; Norbuprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 106.93, 90% CI 2-sided [52.47 to 217.91]
Statistical Analysis 10: Comparison: HCV Without Hepatic Impairment vs No Hepatic Disease or Impairment; Norbuprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 87.10, 90% CI 2-sided [42.74 to 177.50]
Statistical Analysis 11: Comparison: Hepatic Impairment: Child-Pugh A vs HCV Without Hepatic Impairment; Norbuprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 182.98, 90% CI 2-sided [89.79 to 372.89]
Statistical Analysis 12: Comparison: Hepatic Impairment: Child-Pugh B vs HCV Without Hepatic Impairment; Norbuprenorphine; Test type: Superiority or Other; ratio of parameter means, % = 122.77, 90% CI 2-sided [60.24 to 250.19]
Statistical Analysis 13: Comparison: Hepatic Impairment: Child-Pugh A vs No Hepatic Disease or Impairment; Naloxone; Test type: Superiority or Other; ratio of parameter means, % = 69.12, 90% CI 2-sided [33.45 to 142.82]
Statistical Analysis 14: Comparison: Hepatic Impairment: Child-Pugh B vs No Hepatic Disease or Impairment; Naloxone; Test type: Superiority or Other; ratio of parameter means, % = 282.17, 90% CI 2-sided [141.59 to 562.30]
Statistical Analysis 15: Comparison: Hepatic Impairment: Child-Pugh C vs No Hepatic Disease or Impairment; Naloxone; Test type: Superiority or Other; ratio of parameter means, % = 1497.70, 90% CI 2-sided [724.85 to 3094.59]
Statistical Analysis 16: Comparison: HCV Without Hepatic Impairment vs No Hepatic Disease or Impairment; Naloxone; Test type: Superiority or Other; ratio of parameter means, % = 87.64, 90% CI 2-sided [40.30 to 190.59]
Statistical Analysis 17: Comparison: Hepatic Impairment: Child-Pugh A vs HCV Without Hepatic Impairment; Naloxone; Test type: Superiority or Other; ratio of parameter means, % = 78.86, 90% CI 2-sided [34.34 to 181.12]
Statistical Analysis 18: Comparison: Hepatic Impairment: Child-Pugh B vs HCV Without Hepatic Impairment; Naloxone; Test type: Superiority or Other; ratio of parameter means, % = 321.94, 90% CI 2-sided [144.65 to 716.52]
Statistical Analysis 19: Comparison: Hepatic Impairment: Child-Pugh C vs HCV Without Hepatic Impairment; Naloxone; Test type: Superiority or Other; ratio of parameter means, % = 1708.83, 90% CI 2-sided [744.08 to 3924.47]
Statistical Analysis 20: Comparison: Hepatic Impairment: Child-Pugh A vs No Hepatic Disease or Impairment; Naloxone-3-β-D-Glucuronide; Test type: Superiority or Other; ratio of parameter means, % = 84.20, 90% CI 2-sided [60.92 to 116.38]
Statistical Analysis 21: Comparison: Hepatic Impairment: Child-Pugh B vs No Hepatic Disease or Impairment; Naloxone-3-β-D-Glucuronide; Test type: Superiority or Other; ratio of parameter means, % = 110.98, 90% CI 2-sided [82.02 to 150.17]
Statistical Analysis 22: Comparison: Hepatic Impairment: Child-Pugh C vs No Hepatic Disease or Impairment; Naloxone-3-β-D-Glucuronide; Test type: Superiority or Other; ratio of parameter means, % = 81.97, 90% CI 2-sided [60.03 to 111.92]
Statistical Analysis 23: Comparison: HCV Without Hepatic Impairment vs No Hepatic Disease or Impairment; Naloxone-3-β-D-Glucuronide; Test type: Superiority or Other; ratio of parameter means, % = 82.78, 90% CI 2-sided [59.89 to 114.42]
Statistical Analysis 24: Comparison: Hepatic Impairment: Child-Pugh A vs HCV Without Hepatic Impairment; Naloxone-3-β-D-Glucuronide; Test type: Superiority or Other; ratio of parameter means, % = 101.71, 90% CI 2-sided [74.96 to 138.00]
Statistical Analysis 25: Comparison: Hepatic Impairment: Child-Pugh B vs HCV Without Hepatic Impairment; Naloxone-3-β-D-Glucuronide; Test type: Superiority or Other; ratio of parameter means, % = 134.06, 90% CI 2-sided [101.07 to 177.82]
Statistical Analysis 26: Comparison: Hepatic Impairment: Child-Pugh C vs HCV Without Hepatic Impairment; Naloxone-3-β-D-Glucuronide; Test type: Superiority or Other; ratio of parameter means, % = 99.02, 90% CI 2-sided [73.93 to 132.61]

4. Primary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax) of Buprenorphine, Norbuprenorphine, Naloxone and Naloxone-3-β-D-Glucuronide
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Hepatic Impairment: Child-Pugh A | Hepatic Impairment: Child-Pugh B | Hepatic Impairment: Child-Pugh C | HCV Without Hepatic Impairment | No Hepatic Disease or Impairment
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 8
hours
  Buprenorphine | 1.25 [1.00 to 2.00] | 1.50 [0.500 to 2.00] | 1.00 [0.500 to 2.00] | 1.38 [1.00 to 1.50] | 1.75 [1.00 to 3.00]
  Norbuprenorphine | 1.25 [1.00 to 1.25] | 1.25 [1.00 to 36.0] | 0.875 [0.500 to 6.00] | 1.00 [1.00 to 36.0] | 1.00 [1.00 to 2.00]
  Naloxone | 0.875 [0.500 to 1.25] | 0.750 [0.500 to 1.50] | 0.750 [0.250 to 1.25] | 1.00 [0.500 to 1.00] | 1.13 [0.500 to 2.00]
  Naloxone-3-β-D-Glucuronide | 0.500 [0.500 to 1.00] | 0.750 [0.500 to 0.750] | 0.500 [0.500 to 0.767] | 0.750 [0.750 to 1.00] | 0.500 [0.500 to 1.50]

5. Primary Outcome: Time of the Last Measureable Plasma Concentration (Tlast) of Buprenorphine, Norbuprenorphine, Naloxone and Naloxone-3-β-D-Glucuronide
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Hepatic Impairment: Child-Pugh A | Hepatic Impairment: Child-Pugh B | Hepatic Impairment: Child-Pugh C | HCV Without Hepatic Impairment | No Hepatic Disease or Impairment
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 8
hours
  Buprenorphine | 72.0 [48.0 to 96.0] | 120 [72.0 to 168] | 168 [96.0 to 168] | 71.5 [36.0 to 97.0] | 96.0 [36.0 to 144]
  Norbuprenorphine | 144 [72.0 to 168] | 120 [72.0 to 168] | 48.0 [12.0 to 96.0] | 144 [119 to 169] | 156 [120 to 168]
  Naloxone | 10.0 [6.03 to 12.0] | 24.0 [12.0 to 36.0] | 24.0 [24.0 to 48.0] | 10.0 [8.00 to 24.0] | 10.0 [6.00 to 24.0]
  Naloxone-3-β-D-Glucuronide | 24.0 [12.0 to 36.0] | 24.1 [12.0 to 36.0] | 24.0 [12.0 to 36.0] | 36.0 [24.0 to 36.0] | 36.0 [24.0 to 72.0]

6. Primary Outcome: Percentage of Area Under the Concentration-time Curve From Time Zero to Infinity Due to Extrapolation (%AUCextrap) of Buprenorphine, Norbuprenorphine, Naloxone and Naloxone-3-β-D-Glucuronide
Description: Calculated as:
  (AUC0-inf - AUC0-last)/AUC0-inf * 100
  AUC0-inf, apparent body clearance (CL/F), and apparent volume of distribution during terminal phase (Vz/F) would not have been reported if %AUCextrap was > 20%.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of AUC0-inf
Arm/Group | Hepatic Impairment: Child-Pugh A | Hepatic Impairment: Child-Pugh B | Hepatic Impairment: Child-Pugh C | HCV Without Hepatic Impairment | No Hepatic Disease or Impairment
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 8
percentage of AUC0-inf
  Buprenorphine (6,5,5,5,7) | 17.2 (10.8) | 17.1 (6.68) | 14.2 (3.00) | 17.6 (4.96) | 15.5 (5.00)
  Norbuprenorphine (4,6,5,4,4) | 10.2 (8.67) | 24.3 (12.4) | 36.1 (18.0) | 16.5 (3.85) | 13.1 (9.24)
  Naloxone (5,6,5,4,7) | 6.59 (1.86) | 7.48 (6.18) | 1.30 (0.958) | 5.16 (5.01) | 5.31 (2.51)
  Naloxone-3-β-D-Glucuronide (5,7,6,5,4) | 4.98 (1.74) | 3.34 (1.53) | 3.50 (2.08) | 6.04 (3.60) | 5.13 (3.55)

7. Primary Outcome: Terminal Phase Elimination Rate-Constant (λz) of Buprenorphine, Norbuprenorphine, Naloxone and Naloxone-3-β-D-Glucuronide
Description: For the determination of λz, only those data points judged to describe the terminal log-linear decline resulting in an adjusted coefficient of determination value (R2) > 0.7 were used in the regression. A minimum of 3 data points were used in calculating λz.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | Hepatic Impairment: Child-Pugh A | Hepatic Impairment: Child-Pugh B | Hepatic Impairment: Child-Pugh C | HCV Without Hepatic Impairment | No Hepatic Disease or Impairment
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 8
1/hour
  Buprenorphine (6,5,5,5,7) | 0.0221 (46.0) | 0.0142 (41.0) | 0.0123 (29.5) | 0.0197 (32.6) | 0.0193 (50.2)
  Norbuprenorphine (4,6,5,4,4) | 0.0168 (39.4) | 0.0131 (21.5) | 0.0189 (37.4) | 0.0135 (7.37) | 0.0167 (36.0)
  Naloxone (5,6,5,4,7) | 0.322 (23.0) | 0.127 (53.6) | 0.151 (28.2) | 0.371 (35.6) | 0.337 (35.6)
  Naloxone-3-β-D-Glucuronide (5,7,6,5,4) | 0.0974 (26.0) | 0.117 (32.5) | 0.152 (40.4) | 0.0637 (41.9) | 0.0937 (69.4)

8. Primary Outcome: Terminal Elimination Half-life (t1/2) of Buprenorphine, Norbuprenorphine, Naloxone and Naloxone-3-β-D-Glucuronide
Description: Terminal elimination half-life, calculated as ln(2)/λz. The terminal phase elimination half-life was calculated over a period of at least 2 half-lives.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Hepatic Impairment: Child-Pugh A | Hepatic Impairment: Child-Pugh B | Hepatic Impairment: Child-Pugh C | HCV Without Hepatic Impairment | No Hepatic Disease or Impairment
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 8
hours
  Buprenorphine (6,5,5,5,7) | 31.4 (46.0) | 48.7 (41.0) | 56.4 (29.5) | 35.2 (32.6) | 36.0 (50.2)
  Norbuprenorphine (4,6,5,4,4) | 41.3 (39.4) | 52.9 (21.5) | 36.7 (37.4) | 51.2 (7.37) | 41.4 (36.0)
  Naloxone (5,6,5,4,7) | 2.15 (23.0) | 5.45 (53.6) | 4.58 (28.2) | 1.87 (35.6) | 2.06 (35.6)
  Naloxone-3-β-D-Glucuronide (5,7,6,5,4) | 7.12 (26.0) | 5.91 (32.5) | 4.55 (40.4) | 10.9 (41.9) | 7.40 (69.4)

9. Primary Outcome: Apparent Body Clearance (CL/F) of Buprenorphine and Naloxone
Description: Apparent body clearance (only for buprenorphine and naloxone), calculated as Dose/AUC0-inf.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Hepatic Impairment: Child-Pugh A | Hepatic Impairment: Child-Pugh B | Hepatic Impairment: Child-Pugh C | HCV Without Hepatic Impairment | No Hepatic Disease or Impairment
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 8
L/hr
  Buprenorphine (5,4,5,3,6) | 182 (30.8) | 106 (58.4) | 78.3 (44.6) | 232 (22.6) | 193 (56.0)
  Naloxone (5,6,5,4,7) | 7448 (18.7) | 1824 (195) | 344 (57.0) | 5874 (57.0) | 5148 (53.4)

10. Primary Outcome: Apparent Volume of Distribution During Terminal Phase (Vz/F) of Buprenorphine and Naloxone
Description: Apparent volume of distribution during terminal phase (only for buprenorphine and naloxone), calculated as Dose/(λz • AUC0-inf).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Hepatic Impairment: Child-Pugh A | Hepatic Impairment: Child-Pugh B | Hepatic Impairment: Child-Pugh C | HCV Without Hepatic Impairment | No Hepatic Disease or Impairment
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 8
Liters
  Buprenorphine (5,4,5,3,6) | 7226 (26.1) | 6959 (42.6) | 6373 (28.9) | 9580 (29.1) | 9176 (21.9)
  Naloxone (5,6,5,4,7) | 23150 (28.1) | 14353 (187) | 2272 (66.7) | 15845 (97.9) | 15294 (42.8)

ADVERSE EVENTS:
Time Frame: Days 1 - 21
Arm/Group | Hepatic Impairment: Child-Pugh A | Hepatic Impairment: Child-Pugh B | Hepatic Impairment: Child-Pugh C | HCV Without Hepatic Impairment | No Hepatic Disease or Impairment
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8 | 0/8 | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 8/9 | 7/8 | 6/8 | 10/10 | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hepatic Impairment: Child-Pugh A (N=9) | Hepatic Impairment: Child-Pugh B (N=8) | Hepatic Impairment: Child-Pugh C (N=8) | HCV Without Hepatic Impairment (N=10) | No Hepatic Disease or Impairment (N=8)
Dizziness (Nervous system disorders) | 5 | 2 | 4 | 4 | 5
Somnolence (Nervous system disorders) | 3 | 1 | 1 | 1 | 3
Headache (Nervous system disorders) | 1 | 2 | 0 | 2 | 0
Dysarthria (Nervous system disorders) | 1 | 1 | 1 | 0 | 1
Dizziness postural (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Asterixis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Hypersomnia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Mental impairment (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Sedation (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 1 | 0 | 5 | 3
Nausea (Gastrointestinal disorders) | 5 | 2 | 0 | 2 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 3 | 2 | 2 | 3
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 5 | 3
Chills (General disorders) | 1 | 1 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1 | 4 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Euphoric mood (Psychiatric disorders) | 1 | 2 | 4 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days